CLINICAL TRIAL: NCT05484037
Title: Evaluating a Tele-asthma Self-management Intervention, Canadian Asthma Text Messaging Study (CANATEXTS), Among Adults With Asthma
Brief Title: Application of Telehealth Technology in Asthma Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H21-02767
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Asthma Exacerbation; Quality of Life; Medication Adherence
Keywords: Telehealth; Asthma; Self-management; Asthma action plan; Text messaging; Asthma exacerbation; Randomized controlled; Cost-effectiveness
MeSH Terms: conditions — Medication Adherence; Asthma

STUDY DESIGN:
Intervention Model Description: Will be added later
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research coordinator (RC) and certified respiratory educators (CRE) are unblinded. The main investigator and an independent clinical coordinator will be blinded and collected data for primary and secondary outcomes. Statistician and economic evaluator will be blinded to the study randomized orientation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group/telehealth Arm: will be provided access to their electronic asthma action plan (eAAP) via a web Uniform Resource Locator (URL), receive weekly short message service (SMS) check-ins for one year, and be able to communicate with the site's research coordinator (RC) and Certified Respiratory Educator (CRE) via an integrated and interactive (two-way) SMS feature to manage their asthma
  Interventions: Other: CANATEXTS
- Control group (Active Comparator): Control group/standard care Arm: will receive their written Asthma Action Plan (wAAP) and information on how to use it by the site's Certified Respiratory Educator to manage their asthma
  Interventions: Other: CANATEXTS

INTERVENTIONS:
Other: CANATEXTS — Canadian Asthma Text Messaging (CANATEXTS) is a TH intervention facilitating access to an electronic AAP (eAAP) via a mobile device.
  Other Names: Telehealth intervention

SUMMARY:
Background: While effective treatments are available, asthma control is sub-optimal for many asthma patients. To help patients self-manage their asthma symptoms, provision of an asthma action plan (AAP) in written format (wAAP), with instructions on managing worsening asthma symptoms is recommended, as a standard of care; however, only about half of patients correctly adhere to their AAP. Canadian Asthma Text Messaging Study (CANATEXTS) is a Telehealth (TH) intervention facilitating access to an electronic AAP (eAAP) via a mobile device. In a feasibility study to assess the safety and efficacy of CANATEXTS, an 18% reduction in the relative risk of exacerbation was observed among the intervention group compared to control group. This study will assess the effectiveness of CANATEXTS on asthma outcomes in a Canada-wide study.

Methods: This is a superiority a 2-arm, multi-site randomized control trial (RCT). This study aims to determine if CANATEXTS reduces asthma exacerbation over a 12-month period, improves asthma control, quality of life (QoL) and medication adherence, and is cost-effective. The intervention includes access to an electronic asthma action plan (eAAP) on patients' mobile devices, disease-related education, and weekly reminders via a Short messaging system (SMS) interface. The study will include 620 adult participants with asthma recruited from 14 respiratory clinics across Canada. Participants will be randomly assigned to either Intervention group (eAAP) or Control groups (wAAP). All outcomes of interest will be assessed during three in-person assessments (baseline, 6-month, and 12-month) and two telephone follow-ups (3-month and 9-month). Data will be analyzed with a linear mixed-effects model across all time points. Discussion: TH has the potential to improve adult individuals with asthma's engagement in self-management practices. Our feasibility study showed TH could yield a reduction in asthma exacerbation. If the proposed TH intervention is found to be effective for asthma management in a nation-wide trial, it will generate evidence to support integration of TH in asthma self-management. This study will also provide important information on the cost-effectiveness of CANATEXTS when compared to standard asthma care.

DETAILED DESCRIPTION:
While effective treatment is available, asthma control is sub-optimal for 53% of Canadian patients, mainly due to a lack of adequate communication between the patient and care provider. This especially relates to adherence and inhaler technique. The standard of care for asthma is for a patient to see their physician at their office and ideally includes the physician and/or airways educator giving them an asthma action plan (AAP), normally in written format (wAAP), to help patients self-manage their asthma. The primary goal of wAAP is to facilitate a patient's response to worsening asthma symptoms. The wAAPs have shown to be effective in reducing asthma exacerbation; however, only approximately 50% of patients correctly adhere to it. Recently, Telehealth (TH) has been used to address asthma patients' self-efficacy, disease management, and health outcomes. Although there is increasing use of TH in respiratory medicine, in the absence of a robust evidence base it has been recommended conducting interventions to evaluate the efficacy of TH on asthma outcomes and especially exacerbation. We aim to use a TH technology in developing electronic asthma action plan (eAAP) and evaluate the effectiveness of a telecommunication intervention [(hereafter-called Canadian Asthma Text Messaging Study (CANATEXTS)] on improving asthma outcomes among adult asthma patients. The CANATEXTS intervention will digitalis a patient's wAAP to access and use online, will send patients a weekly text message reminders to complete their asthma diary and assess their level of asthma control. If the asthma control is sub-optimal, guided by their action plan, patients will adjust their therapy. The goal is to improve patient health outcomes via enhancing patient-physician interaction and using a more practical electronic asthma action plan model (eAAP). The Primary objective is to determine the effectiveness of CANATEXTS in reducing exacerbation over a 12-month period. The Secondary objectives are to determine the effectiveness of our intervention on quality of life and asthma control, and medication adherence. The cost-effectiveness of the CANATEXTS intervention for improving asthma outcomes when compared to standard care will also be assessed. Our previous TH feasibility study showed the efficacy of this intervention with asthma patients, in which 92% of participants showed a strong commitment to study completion. In our study, we found that the exacerbation rate was reduced by 18% in the intervention group (eAAP), when compared to the control group (wAAP). In the proposed CANATEXTS study, we endeavour to increase the precision of the intervention effect estimate (to 25%), improve accessibility and usability of CANATEXTS (e.g., engaged patients in the design of the intervention and incorporate their perspectives to improve the TH intervention), and include patients from across Canada. A well-known digital health platform that aims to deliver better care for all (call WelTel technology Platform) will be applied in the study, as it was applied in our feasibility study. We calculated a sample size of 622 asthma patients, which will be recruited from collaborating asthma clinics from multiple sites across Canada, predicting a 25% absolute reduction in exacerbation rates between the two study groups. The study participants will be randomly allocated to two study groups: (1) The intervention group will receive the standard care and have access to their AAP online (eAAP), while receiving weekly text messages (SMS) reminders to check-in their eAAP for 12 months for assessment of their asthma control. They will also be able to send and receive 2-way SMS for their non-emergency queries. (2) The control group will receive the standard care, have access to written-based AAP (wAAP), and education on how to use their wAAP. Both study groups will have access to self-management educational materials and will be treated according to the step-wise approach recommended in the Canadian Asthma Continuum. After subjects provide written informed consent, they will see a certified airways educator to receive an individualized action plan, an appropriate education on how to use their AAP, and will then meet the study coordinator to complete baseline questionnaires documenting their demographics, asthma history (including number of exacerbation within the past 12 months), current asthma control, and work productivity and activity impairment, as well as spirometry test (a pulmonary function test for measuring a patient's lung capacity and breath). We will also assess asthma quality of life, medication adherence, and asthma control using validated measurement tools. Furthermore, we will also assess how confident patients feel in controlling their asthma, using a measure of self-efficacy, attitudes, and knowledge. Study subjects will be seen at 6 and 12 months post initial assessment to assess their asthma control (specifically asthma exacerbation) and the use of health care resources. In addition, we will conduct telephone calls at 3 and 9 months post initial assessment to track health care utilization and exacerbation history. All outcomes of interest will be assessed during the three in-person assessments and the two telephone follow-up calls. A comparison of both groups on primary and secondary outcomes will be made at the end of the trial (month 12) to analyze data based on sex, age, disease severity, disease duration, and education level. Hypothesis: We expect to observe a significant reduction in asthma exacerbation rates among the intervention group (eAAP), when compared to the control group (wAAP). We further hypothesize that the eAAP subjects will have an improvement in secondary measures including quality of life, better asthma control and medication adherence. We believe the CANATEXTS intervention will work more effectively and yield better asthma outcomes in the intervention group, than it did in our feasibility study. We also believe that our proposed TH intervention will be more cost-effective when compared to standard care for asthma management in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis asthma
* Must have history of one exacerbation in the previous year
* Must have moderate or severe asthma
* Must be prescribed both reliever and controller medications
* Must be capable to communicate in English or French
* Mush have a digital device with access to the internet

Exclusion Criteria:

- Patients with chronic obstructive pulmonary disease (COPD)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Yes, based on self-representation of gender identity.
Enrollment: 620 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Exacerbation | Every 6 months up to one year
  An asthma attack that requires either taking a course of Oral Corticosteroids (OCS) for at least three days, or an asthma-related emergency room (ED) visit or hospitalization

SECONDARY OUTCOMES:
Asthma control | Every 6 months up to one year
  How well asthma is under control that will be measured using standard asthma control assessment
Medication adherence | every 6 months up to one year
  Adherence to prescribed medication by taking prescribed medication routinely. Will be measured using standard adherence checklist

OTHER OUTCOMES:
Cost effectiveness | at the end of year 3 through year four of the intervention
  Trade-off between the incremental costs and incremental effectiveness of telehealth technology

CONTACTS AND LOCATIONS:
Overall Officials: Chris Carlsten, M.D., Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Centre for Clinical Epidemiology and Evaluation, Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - The Lung Centre, Vancouver Coastal Health, 7th Floor 2775 Laurel Street, Vancouver, British Columbia
  - University of British Columbia - Vancouver Coastal Health, Vancouver, British Columbia